CLINICAL TRIAL: NCT05741736
Title: Five Days for Health (FDH): Small Group-based Lifestyle Modification Program on Weight Loss
Acronym: FDH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinical Hospital Centre Zagreb (Other)
Collaborators: Croatian Institute of Public Health (Unknown)
Responsible Party: Principal Investigator, Maja Baretić, Specialis of internal medicine, consultant endocriologist and diabetologist, assistant professor, Clinical Hospital Centre Zagreb
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 02/013-JG
Record Dates: First submitted 2023-02-04; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Obesity; Overweight
Keywords: obesity; overweight; lifestyle modification; weight loss; small group program; multidisciplinary team
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group (Other): A structured 5-day lifestyle modification program led by endocrinologists-diabetologists together with a nutritionist, a psychologist, and a kinesiologist is aiming to educate on lifestyle modification necessary to lose weight.
  Interventions: Behavioral: five-days small group-based lifestyle modification program

INTERVENTIONS:
Behavioral: five-days small group-based lifestyle modification program — healthy lifestyle, based on the promotion of a particular dietary pattern, regular physical activity, psychological support, education, and small group intervention results in weight loss

SUMMARY:
Croatia is according to statistical data one of the countries in the European Union with the highest percentages of overweight and obese inhabitants. Since the nature of obesity is multifactorial, a multidisciplinary team should treat it in a comprehensive way. A healthy lifestyle, based on the promotion of a particular dietary pattern, regular physical activity, psychological support, education, and small group intervention results in weight loss. We are aiming to develop a five-days small group-based lifestyle modification program on weight loss that would be appropriate in the general practice and outpatient setting facilities. A structured 5-day lifestyle modification program led by endocrinologists-diabetologists together with a nutritionist, a psychologist, and a kinesiologist is aiming to educate on lifestyle modification necessary to lose weight.

DETAILED DESCRIPTION:
The program involves coherent groups of motivated participants in smaller groups of 7-10 persons. Participants are adults with body mass index (BMI) in the range of overweight or obese and are motivated to change their lifestyle. During the five days of the program held outside the medical facility positive interaction and mutual support of the participants develop in the group together with education and an informal approach, along with practical workshops on nutrition, daily physical activity and psychological support, patients receive practical recommendations for life. Follow-up continues in the form of short additional educational lectures, support, and body weight measurement after one month, three months, six months and after a year. Participants are encouraged to stay in contact between the meetings using the same instant messaging platform in a form of a closed group, and a leader of the program is sending inspirational messages and advice regularly. Initially, after 3 and 6 months a metabolic parameter evaluation is performed (fasting glucose and insulin, lipid profile) as well as blood pressure is measured. Individual anthropometric measurements of the participants are carried out on the first day of the program and continued at every visit. The parameters taken are body height (cm), body mass (kg), waist circumference (cm), hip circumference (cm), BMI (kg/m2), the proportion of fat tissue (%) and muscle tissue (%), basal metabolism (kcal) and visceral adipose tissue. On the first day of the program, an initial questionnaire is filled out exploring sociodemographic and health data, data on eating habits, physical activity and psychological.

Education During the 5-day participants have lectures explaining in a simple short interactive lecture a different topic related to obesity followed by discussion. Topics explain concerns about obesity as a disease, the background of obesity, metabolic and cardiovascular consequences of obesity, nonverbal communication and obesity, the plateau phenomenon and the epidemiology of obesity.

Nutrition The program helps participants to make healthier food choices by acquiring knowledge of nutrition basics and meal planning. During the program, the participants learn how to prepare easy and healthy meals for breakfast, lunch, dinner and snack, read food labels and measure portion sizes with their hands.

Physical activity Participants wear accelerometers before the beginning of the program. During the program, they are going to have daily 10' physical exercises (exercise and explanations) in a form of a complex of exercises designed for all adults, especially for the working population. The set of exercises consists of stretching and mobility exercises that are performed with light, moderate movements and can be performed without hindrance in everyday work clothes. They are going to be educated on how and how much to be physically active and how to choose the appropriate physical activity and activity intensity.

Psychological support Daily support involves behavioural change that is working on goal setting and recognizing the advantages and disadvantages of changing behaviour. Nex workshop works on recognizing the difference between emotional hunger and physical hunger, identifying personal triggers, and finding alternatives to emotional eating. Participants identify the key distortions in the negative thoughts of dieters that prevent them from reaching and maintaining their desired weight and learn how to correct these distortions. Also, they learn what it means to have a positive or negative body image, how body image affects mental and physical health, and what we can do to improve our body image.

Evaluation At the end of each lecture/interactive workshop, participants fill out an evaluation questionnaire. At the end of the education, on the 5th day of education, the participants fille out the final questionnaire (outcome evaluation).

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants between the ages of 18 and 70
* body mass index (BMI kg/m2) between 25-45
* able to travel regularly to the study location
* interested in participating in a weight loss program.

Exclusion Criteria:

* currently enrolled in another organized weight loss program
* taking medications that affect appetite (unless dosage had been stable for at least the previous six months)
* history of gastric bypass or other surgical weight loss procedures
* medical conditions (e.g., cancer, substance abuse, psychotic disorders) that could limit their ability to comply with the behavioral recommendations or pose a risk to the participant during weight loss
* pregnancy or planning to become pregnant during the next two years -
* breastfeeding
* consuming an amount of alcohol that could interfere with study completion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-01-23 (Actual); Primary Completion 2024-12-23 (Estimated); Study Completion 2024-12-23 (Estimated)

PRIMARY OUTCOMES:
weight loss | 12 months
  difference between basal weight and after 12 months

SECONDARY OUTCOMES:
body composition | 12 months
  difference between basal fat percentage and after 12 months
metabolic parameters | 12 months
  difference between basal fasting glucose and lipid profila and after 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Maja Baretić, Principal Investigator — Clinical Hospital Centre Zagreb
Locations (2):
- Croatia (2):
  - Croatian Institute of Public Health, Zagreb
  - Universtiy Hospital Centre Zagreb, Zagreb

IPD SHARING:
Plan to Share IPD: No
on request